CLINICAL TRIAL: NCT05566340
Title: Surgical Treatment of Aortic Valve Disease With Moderate Functional Mitral Regurgitation
Brief Title: Treatment of Moderate FMR During AVR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fuwai Yunnan Cardiovascular Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FZX2019-06-01 2022YFKY088
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Functional Mitral Regurgitation
Keywords: functional mitral regurgitation; aortic valve replacement; mitral valve repair
MeSH Terms: interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- isolated aortic valve replacement group: Isolated aortic valve replacement surgery.
  Interventions: Procedure: mitral valve repair
- aortic valve replacement with mitral valve repair group: Aortic valve replacement with mitral valve repair
  Interventions: Procedure: mitral valve repair

INTERVENTIONS:
Procedure: mitral valve repair — Repair of mitral valve concomitant to aortic valve replacement.

SUMMARY:
Debates exist on the treatment of moderate functional mitral regurgitation (FMR) in patients undergoing aortic valve replacement (AVR) for aortic valve disease. This study aims to evaluate the left ventricular function, which was evaluated through global longitudinal strain, after isolated AVR and AVR + mitral valve repair (MVr) in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received AVR (with or without concomitant MVr) from two center (Fuwai Yunnan Cardiovascular Hospital and Fuwai Hospital, Chinese Academy of Medical Sciences).
2. Age more than 18 years.

Exclusion Criteria:

1. Those with a history of rheumatic valvular disease or infective endocarditis.
2. Primary mitral valve lesions.
3. Patients receiving mitral valve replacement.
4. Patient who refuse to participate in this study, or cannot complete 6-month follow-up after surgery.
5. Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 154 patients with moderate FMR undergoing isolated AVR or AVR + MVr will be prospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
left ventricular global longitudinal strain | 10/10/2022-10/10/2023
  The change of left ventricular global longitudinal strain compared to before surgery

IPD SHARING:
Plan to Share IPD: No